CLINICAL TRIAL: NCT00583531
Title: A Pilot Study of the Safety and Efficacy of AST-120 in the Treatment of Antibiotic-Refractory Pouchitis
Brief Title: Safety and Efficacy of AST-120 in the Treatment of Antibiotic-Refractory Pouchitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Ocera Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-007216
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Pouchitis
Keywords: Antibiotic-refractory Pouchitis; Pouchitis; Ulcerative Colitis
MeSH Terms: conditions — Pouchitis; Colitis, Ulcerative | interventions — AST 120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): Active treatment with AST-120
  Interventions: Drug: AST-120

INTERVENTIONS:
Drug: AST-120 — Oral, 2 grams TID in sachets for 4 weeks

SUMMARY:
This is an open-label pilot study in which all patients will receive AST-120 for 4 weeks. Patients will discontinue antibiotics at study entry. They may continue other previously prescribed treatments (e.g., probiotics and/or nutritional agents) at the discretion of the study doctor. The purpose of the study is to assess whether the investigational medication AST-120 will be a safe and effective treatment for the symptoms of pouchitis, a chronic inflammatory condition, in patients whose symptoms have not responded well to antibiotics. An initial group of 10 patients will be enrolled. If there are no serious side effects associated with the study drug and at least 3 of the 10 patients respond, a second group of 10 patients may be enrolled. Patients will have clinic visits at the start of the study and at week 4. Patients will be checked by phone on a weekly basis for symptom response, compliance and development of side effects. Endoscopies will be performed at the start of the study and at week 4 or early termination.

DETAILED DESCRIPTION:
Patients with acute pouchitis are typically treated with metronidazole or ciprofloxacin for 10-14 days. Most patients with pouchitis respond to these or other antibiotics. Patients who experience frequent relapses and those with chronic pouchitis will require long term maintenance antibiotics. Probiotics may be considered as an alternate to chronic antibiotic therapy for maintenance of remission in chronic antibiotic-dependent pouchitis. In practice, we would institute maintenance therapy for patients who relapse at least 3 times within one year, or within 1 month of discontinuation of antibiotics. Among patients receiving maintenance antibiotics who develop loss of clinical benefit after prolonged treatment, rotation of three or four antibiotics in 1-week intervals may be beneficial. Patients who do not improve with single antibiotics may respond to combination therapy with two antibiotics. If not, they can be treated with topical or oral budesonide. Other options include topical mesalamine (enemas or suppositories), oral sulfasalazine or mesalamine, other topical or oral steroids, and possibly oral bismuth, azathioprine, 6-mercaptopurine or infliximab. However, there is little evidence base for these therapies in the literature, and many of these therapies are expensive and/or potentially toxic. A therapy that does not suppress the immune system, and that has little or no toxicity would be attractive for patients with antibiotic-refractory pouchitis.

AST-120 is manufactured by Kureha Corporation, Japan. The agent was approved in Japan in 1991 for the treatment of patients with chronic kidney disease(CKD). It is comprised of highly adsorptive, porous, spherical carbon particles and is packaged in 2 g sachets for oral administration designed for the treatment of gastrointestinal diseases. AST-120 consists of black microspheres approximately 0.2-0.4 mm in diameter with high adsorption ability and large surface area. Composed mainly of carbon (approximately 96%), the clinical utility of AST-120 is thought to reside in its ability to adsorb small molecular weight toxins, inflammatory mediators, and harmful bile acid products from the gastrointestinal tract, preventing local toxicity and their systemic absorption. AST-120 has a selective adsorption profile for certain acidic and basic organic compounds, and has a significantly lower adsorptive capacity than activated charcoal for digestive enzymes.

In this study, patients with active pouchitis after ileal pouch-anal anastomosis (IPAA) for Ulcerative Colitis with primary symptoms such as increased stool frequency and abdominal pain, and refractory to antibiotics (do not respond to antibiotic therapy for a minimum of 14 days) will be enrolled. Patients must have active pouchitis confirmed by endoscopy and biopsy within 4 weeks of study entry. The diagnosis of active pouchitis will be defined by a PDAI score >7 points, with a combined assessment of symptoms, endoscopy and histology.

Eligible patients will receive AST-120 sachets at 2g three times daily (TID) to be taken between meals at 10:00 am, 3:00 pm and immediately before going to bed for 4 complete weeks. AST-120 is a tasteless, odorless, oral preparation. To take the product, patients will tear open the sachets, drop the contents directly on their tongue and wash it down with 8 ounces of water. Patients will be evaluated at baseline and week 4 or early termination by the study physician, including endoscopies with histology and routine laboratory tests. Patients will be checked on a weekly basis by the study coordinator by phone for symptom response, compliance, and development of adverse events. Quality of Life Assessments (Cleveland Global Quality of Life and Short Inflammatory Bowel Questionnaire) will be conducted at baseline and week 4 or early termination. A patient is defined as having completed study treatment if he/she has received investigational product and is followed for safety through the last on-site visit of the 4 week treatment course.

Any co-prescribed medicine must be given at least 30 minutes before AST-120 administration. The following drugs for pouchitis can be co-prescribed/maintained during AST-120 treatment and their utilization will be recorded as secondary endpoints:

* Antidiarrheal therapy with loperamide (Imodium)
* Nutritional agents and Probiotics at the same dose as previously prescribed, if the dose has been stable for 2 weeks at study entry.

Antibiotics must be stopped by the time of entry into the study. However, antibiotics prescribed to treat infection other than pouchitis will be allowed and recorded.

The need to prescribe any of the following drugs during the study will constitute treatment failure:

* Oral or topical corticosteroids
* Oral or topical 5-ASA
* Nutritional agents (SCFA enemas or suppositories, glutamine, dietary fibers)
* Probiotics
* Narcotic-based antidiarrheal agents

In addition patients will be considered to have failed treatment if they have a PDAI score improvement of < or = 2 points at the end of the trial. Patients will be discontinued from the study if they become pregnant or if warranted by treatment-emergent safety concerns or if, in the opinion of the investigator, it is in the patient's best interest to discontinue the study.

A first cohort of 10 patients will be treated; based on outcome (efficacy and safety: no significant Adverse Event (AE) associated with study drug and at least 3/10 patients responding) a second cohort of 10 patients may be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active pouchitis (defined as having a PDAI score > 7) after IPAA for UC, despite at least 14 days of antibiotic therapy. Active pouchitis must be confirmed by endoscopy and histology within 4 weeks of study entry
* Able to give informed consent
* Able and willing to comply with all study procedures

Exclusion Criteria:

* Patients previously treated with infliximab or any investigational immunosuppressant/ immunomodulator for pouchitis
* Patients undergoing chemotherapy for the treatment of cancer
* Presence of other inflammatory diseases of the pouch: Crohn's disease, Cuffitis, active specific infection of the pouch: (e.g., CMV, C. difficile)
* History of non-inflammatory disease of the pouch: decreased pouch compliance, irritable pouch syndrome, afferent or efferent limb obstruction, stricture of pouch
* Ileal pouch patients with familial adenomatous polyposis
* History of other diarrheal illnesses: lactose intolerance, celiac disease, small bowel bacterial overgrowth
* Primary Sclerosing Cholangitis with or without liver transplant
* Uncontrolled systemic disease
* Needing oral or topical 5-ASA, cholestyramine, steroids or immunomodulators
* Other major physical or major psychiatric illness within the last 6 months that in the opinion of the investigator would affect the patient's ability to complete the trial
* Women who are pregnant, breast feeding, or planning to become pregnant during the study
* Women of child-bearing potential who are not willing to use barrier or depot contraception methods
* Use of NSAIDs or aspirin (>3 times per week) within the past 3 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Response as defined by a decrease in the Pouchitis Diseases Activity Index (PDAI) score of at least 3 points | 4 weeks
Safety: Any adverse events (AEs) deemed possibly, probably, or definitely related to treatment with investigational product during 4 weeks of treatment | 4 weeks

SECONDARY OUTCOMES:
Remission, as defined as a PDAI score of less than 7 points | 4 weeks
Reduction of PDAI clinical symptom subscore of at least 1 point | 4 weeks
Reduction of PDAI endoscopic subscore of at least 1 point | 4 weeks
Reduction of PDAI histology subscore of at least 1 point | 4 weeks
Need for rescue medication/quantity of antidiarrheal medication used during the last week of the trail compared to usage in the week prior to study entry | 4 weeks
Quality of Life as measured by the Cleveland Global QoL instrument and Short Inflammatory Bowel Disease Questionnaire (SIBDQ) | 4 weeks
Significant change in clinical laboratory tests | 4 weeks
Worsening GI symptoms (diarrhea, abdominal pain, urgency or bleeding) or new GI and extra-GI symptoms (e.g., headache, nausea, vomiting, constipation) | 4 weeks
Significant change in physical examination, including vital signs (blood pressure, heart rate, respiration rate and temperature) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Darrell S. Pardi, MD, Principal Investigator — Mayo Clinic College of Medicine
Locations (1):
- Mayo Clinic, Inflammatory Bowel Disease Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Sandborn WJ. Pouchitis following ileal pouch-anal anastomosis: definition, pathogenesis, and treatment. Gastroenterology. 1994 Dec;107(6):1856-60. doi: 10.1016/0016-5085(94)90832-x. No abstract available. PMID 7958702
- [Background] Fazio VW, Ziv Y, Church JM, Oakley JR, Lavery IC, Milsom JW, Schroeder TK. Ileal pouch-anal anastomoses complications and function in 1005 patients. Ann Surg. 1995 Aug;222(2):120-7. doi: 10.1097/00000658-199508000-00003. PMID 7639579
- [Background] Simchuk EJ, Thirlby RC. Risk factors and true incidence of pouchitis in patients after ileal pouch-anal anastomoses. World J Surg. 2000 Jul;24(7):851-6. doi: 10.1007/s002680010136. PMID 10833254
- [Background] Salemans JM, Nagengast FM, Lubbers EJ, Kuijpers JH. Postoperative and long-term results of ileal pouch-anal anastomosis for ulcerative colitis and familial polyposis coli. Dig Dis Sci. 1992 Dec;37(12):1882-9. doi: 10.1007/BF01308083. PMID 1335407
- [Background] Marcello PW, Roberts PL, Schoetz DJ Jr, Coller JA, Murray JJ, Veidenheimer MC. Long-term results of the ileoanal pouch procedure. Arch Surg. 1993 May;128(5):500-3; discussion 503-4. doi: 10.1001/archsurg.1993.01420170030003. PMID 8489382
- [Background] Meagher AP, Farouk R, Dozois RR, Kelly KA, Pemberton JH. J ileal pouch-anal anastomosis for chronic ulcerative colitis: complications and long-term outcome in 1310 patients. Br J Surg. 1998 Jun;85(6):800-3. doi: 10.1046/j.1365-2168.1998.00689.x. PMID 9667712
- [Background] Svaninger G, Nordgren S, Oresland T, Hulten L. Incidence and characteristics of pouchitis in the Kock continent ileostomy and the pelvic pouch. Scand J Gastroenterol. 1993 Aug;28(8):695-700. doi: 10.3109/00365529309098275. PMID 8210985
- [Background] Shepherd NA, Hulten L, Tytgat GN, Nicholls RJ, Nasmyth DG, Hill MJ, Fernandez F, Gertner DJ, Rampton DS, Hill MJ, et al. Pouchitis. Int J Colorectal Dis. 1989 Dec;4(4):205-29. doi: 10.1007/BF01644986. No abstract available. PMID 2693561
- [Background] Sandborn WJ. Pouchitis: risk factors, frequency, natural history, classification and public health perspective. Kluwer Academic Publishers, 1997.
- [Background] Sandborn WJ, Pardi DS. Clinical management of pouchitis. Gastroenterology. 2004 Dec;127(6):1809-14. doi: 10.1053/j.gastro.2004.10.011. No abstract available. PMID 15578518
- [Background] Sagar PM, Pemberton JH. Ileo-anal pouch function and dysfunction. Dig Dis. 1997 May-Jun;15(3):172-88. doi: 10.1159/000171597. PMID 9158926
- [Background] Lohmuller JL, Pemberton JH, Dozois RR, Ilstrup D, van Heerden J. Pouchitis and extraintestinal manifestations of inflammatory bowel disease after ileal pouch-anal anastomosis. Ann Surg. 1990 May;211(5):622-7; discussion 627-9. PMID 2339922
- [Background] Tytgat GN, van Deventer SJ. Pouchitis. Int J Colorectal Dis. 1988 Nov;3(4):226-8. doi: 10.1007/BF01660720. No abstract available. PMID 3058838
- [Background] Shen B, Achkar JP, Lashner BA, Ormsby AH, Remzi FH, Bevins CL, Brzezinski A, Petras RE, Fazio VW. Endoscopic and histologic evaluation together with symptom assessment are required to diagnose pouchitis. Gastroenterology. 2001 Aug;121(2):261-7. doi: 10.1053/gast.2001.26290. PMID 11487535
- [Background] Hurst RD, Molinari M, Chung TP, Rubin M, Michelassi F. Prospective study of the incidence, timing and treatment of pouchitis in 104 consecutive patients after restorative proctocolectomy. Arch Surg. 1996 May;131(5):497-500; discussion 501-2. doi: 10.1001/archsurg.1996.01430170043007. PMID 8624195
- [Background] Duffy M, O'Mahony L, Coffey JC, Collins JK, Shanahan F, Redmond HP, Kirwan WO. Sulfate-reducing bacteria colonize pouches formed for ulcerative colitis but not for familial adenomatous polyposis. Dis Colon Rectum. 2002 Mar;45(3):384-8. doi: 10.1007/s10350-004-6187-z. PMID 12068199
- [Background] Gosselink MP, Schouten WR, van Lieshout LM, Hop WC, Laman JD, Ruseler-van Embden JG. Eradication of pathogenic bacteria and restoration of normal pouch flora: comparison of metronidazole and ciprofloxacin in the treatment of pouchitis. Dis Colon Rectum. 2004 Sep;47(9):1519-25. doi: 10.1007/s10350-004-0623-y. Epub 2004 Jul 8. PMID 15486751
- [Background] Gionchetti P, Rizzello F, Venturi A, Ugolini F, Rossi M, Brigidi P, Johansson R, Ferrieri A, Poggioli G, Campieri M. Antibiotic combination therapy in patients with chronic, treatment-resistant pouchitis. Aliment Pharmacol Ther. 1999 Jun;13(6):713-8. doi: 10.1046/j.1365-2036.1999.00553.x. PMID 10383499
- [Background] Kmiot WA, Youngs D, Tudor R, Thompson H, Keighley MR. Mucosal morphology, cell proliferation and faecal bacteriology in acute pouchitis. Br J Surg. 1993 Nov;80(11):1445-9. doi: 10.1002/bjs.1800801132. PMID 8252361
- [Background] Nasmyth DG, Godwin PG, Dixon MF, Williams NS, Johnston D. Ileal ecology after pouch-anal anastomosis or ileostomy. A study of mucosal morphology, fecal bacteriology, fecal volatile fatty acids, and their interrelationship. Gastroenterology. 1989 Mar;96(3):817-24. PMID 2914643
- [Background] Schmidt CM, Lazenby AJ, Hendrickson RJ, Sitzmann JV. Preoperative terminal ileal and colonic resection histopathology predicts risk of pouchitis in patients after ileoanal pull-through procedure. Ann Surg. 1998 May;227(5):654-62; discussion 663-5. doi: 10.1097/00000658-199805000-00006. PMID 9605657
- [Background] Stahlberg D, Gullberg K, Liljeqvist L, Hellers G, Lofberg R. Pouchitis following pelvic pouch operation for ulcerative colitis. Incidence, cumulative risk, and risk factors. Dis Colon Rectum. 1996 Sep;39(9):1012-8. doi: 10.1007/BF02054692. PMID 8797652
- [Background] Hata K, Watanabe T, Shinozaki M, Nagawa H. Patients with extraintestinal manifestations have a higher risk of developing pouchitis in ulcerative colitis: multivariate analysis. Scand J Gastroenterol. 2003 Oct;38(10):1055-8. doi: 10.1080/00365520310005938. PMID 14621280
- [Background] Penna C, Dozois R, Tremaine W, Sandborn W, LaRusso N, Schleck C, Ilstrup D. Pouchitis after ileal pouch-anal anastomosis for ulcerative colitis occurs with increased frequency in patients with associated primary sclerosing cholangitis. Gut. 1996 Feb;38(2):234-9. doi: 10.1136/gut.38.2.234. PMID 8801203
- [Background] Achkar JP, Al-Haddad M, Lashner B, Remzi FH, Brzezinski A, Shen B, Khandwala F, Fazio V. Differentiating risk factors for acute and chronic pouchitis. Clin Gastroenterol Hepatol. 2005 Jan;3(1):60-6. doi: 10.1016/s1542-3565(04)00604-4. PMID 15645406
- [Background] Shen B, Fazio VW, Remzi FH, Delaney CP, Bennett AE, Achkar JP, Brzezinski A, Khandwala F, Liu W, Bambrick ML, Bast J, Lashner B. Comprehensive evaluation of inflammatory and noninflammatory sequelae of ileal pouch-anal anastomoses. Am J Gastroenterol. 2005 Jan;100(1):93-101. doi: 10.1111/j.1572-0241.2005.40778.x. PMID 15654787
- [Background] Sandborn WJ, Landers CJ, Tremaine WJ, Targan SR. Antineutrophil cytoplasmic antibody correlates with chronic pouchitis after ileal pouch-anal anastomosis. Am J Gastroenterol. 1995 May;90(5):740-7. PMID 7733080
- [Background] Aisenberg J, Legnani PE, Nilubol N, Cobrin GM, Ellozy SH, Hegazi RA, Yager J, Bodian C, Gorfine SR, Bauer JJ, Plevy SE, Sachar DB. Are pANCA, ASCA, or cytokine gene polymorphisms associated with pouchitis? Long-term follow-up in 102 ulcerative colitis patients. Am J Gastroenterol. 2004 Mar;99(3):432-41. doi: 10.1111/j.1572-0241.2004.04107.x. PMID 15056081
- [Background] Merrett MN, Mortensen N, Kettlewell M, Jewell DO. Smoking may prevent pouchitis in patients with restorative proctocolectomy for ulcerative colitis. Gut. 1996 Mar;38(3):362-4. doi: 10.1136/gut.38.3.362. PMID 8675087
- [Background] Di Febo G, Miglioli M, Lauri A, Biasco G, Paganelli GM, Poggioli G, Gozzetti G, Barbara L. Endoscopic assessment of acute inflammation of the ileal reservoir after restorative ileo-anal anastomosis. Gastrointest Endosc. 1990 Jan-Feb;36(1):6-9. doi: 10.1016/s0016-5107(90)70912-1. PMID 2155847
- [Background] Moskowitz RL, Shepherd NA, Nicholls RJ. An assessment of inflammation in the reservoir after restorative proctocolectomy with ileoanal ileal reservoir. Int J Colorectal Dis. 1986 Jul;1(3):167-74. doi: 10.1007/BF01648445. PMID 3039030
- [Background] Shen B, Shermock KM, Fazio VW, Achkar JP, Brzezinski A, Bevins CL, Bambrick ML, Remzi FH, Lashner BA. A cost-effectiveness analysis of diagnostic strategies for symptomatic patients with ileal pouch-anal anastomosis. Am J Gastroenterol. 2003 Nov;98(11):2460-7. doi: 10.1111/j.1572-0241.2003.07710.x. PMID 14638349
- [Background] Shepherd NA, Jass JR, Duval I, Moskowitz RL, Nicholls RJ, Morson BC. Restorative proctocolectomy with ileal reservoir: pathological and histochemical study of mucosal biopsy specimens. J Clin Pathol. 1987 Jun;40(6):601-7. doi: 10.1136/jcp.40.6.601. PMID 3611389
- [Background] Parsi MA, Shen B, Achkar JP, Remzi FF, Goldblum JR, Boone J, Lin D, Connor JT, Fazio VW, Lashner BA. Fecal lactoferrin for diagnosis of symptomatic patients with ileal pouch-anal anastomosis. Gastroenterology. 2004 May;126(5):1280-6. doi: 10.1053/j.gastro.2004.02.012. PMID 15131788
- [Background] Johnson MW, Dewar DH, Ciclitira P, Forbes A, Nicholls RJ, Bjarnason I. Use of fecal lactoferrin to diagnose irritable pouch syndrome: a word of caution. Gastroenterology. 2004 Nov;127(5):1647-8; author reply 1648. doi: 10.1053/j.gastro.2004.09.069. No abstract available. PMID 15521043
- [Background] Mann SD, Pitt J, Springall RG, Thillainayagam AV. Clostridium difficile infection--an unusual cause of refractory pouchitis: report of a case. Dis Colon Rectum. 2003 Feb;46(2):267-70. doi: 10.1007/s10350-004-6533-1. PMID 12576902
- [Background] Seggerman RE, Chen MY, Waters GS, Ott DJ. Pictorial essay. Radiology of ileal pouch-anal anastomosis surgery. AJR Am J Roentgenol. 2003 Apr;180(4):999-1002. doi: 10.2214/ajr.180.4.1800999. No abstract available. PMID 12646444
- [Background] Libicher M, Scharf J, Wunsch A, Stern J, Dux M, Kauffmann GW. MRI of pouch-related fistulas in ulcerative colitis after restorative proctocolectomy. J Comput Assist Tomogr. 1998 Jul-Aug;22(4):664-8. doi: 10.1097/00004728-199807000-00029. PMID 9676464
- [Background] Shen B, Lashner BA, Bennett AE, Remzi FH, Brzezinski A, Achkar JP, Bast J, Bambrick ML, Fazio VW. Treatment of rectal cuff inflammation (cuffitis) in patients with ulcerative colitis following restorative proctocolectomy and ileal pouch-anal anastomosis. Am J Gastroenterol. 2004 Aug;99(8):1527-31. doi: 10.1111/j.1572-0241.2004.30518.x. PMID 15307872
- [Background] Thompson-Fawcett MW, Mortensen NJ, Warren BF. "Cuffitis" and inflammatory changes in the columnar cuff, anal transitional zone, and ileal reservoir after stapled pouch-anal anastomosis. Dis Colon Rectum. 1999 Mar;42(3):348-55. doi: 10.1007/BF02236352. PMID 10223755
- [Background] Keighley MR. Review article: the management of pouchitis. Aliment Pharmacol Ther. 1996 Aug;10(4):449-57. doi: 10.1046/j.1365-2036.1996.32174000.x. PMID 8853749
- [Background] Munoz-Juarez M, Pemberton JH, Sandborn WJ, Tremaine WJ, Dozois RR. Misdiagnosis of specific cytomegalovirus infection of the ileoanal pouch as refractory idiopathic chronic pouchitis: report of two cases. Dis Colon Rectum. 1999 Jan;42(1):117-20. doi: 10.1007/BF02235196. PMID 10211531
- [Background] Moonka D, Furth EE, MacDermott RP, Lichtenstein GR. Pouchitis associated with primary cytomegalovirus infection. Am J Gastroenterol. 1998 Feb;93(2):264-6. doi: 10.1111/j.1572-0241.1998.00264.x. PMID 9468256
- [Background] Salfiti N, Loftus EV, Tremaine WJ, Pardi DS, et al. Clinical features and outcomes of cytomegalovirus colitis or pouchitis in patients with inflammatory bowel disease. Am J Gastroenterol 100:S316, 2005
- [Background] Shen B, Achkar JP, Lashner BA, Ormsby AH, Brzezinski A, Soffer EE, Remzi FH, Bevins CL, Fazio VW. Irritable pouch syndrome: a new category of diagnosis for symptomatic patients with ileal pouch-anal anastomosis. Am J Gastroenterol. 2002 Apr;97(4):972-7. doi: 10.1111/j.1572-0241.2002.05617.x. PMID 12003434
- [Background] Prudhomme M, Dozois RR, Godlewski G, Mathison S, Fabbro-Peray P. Anal canal strictures after ileal pouch-anal anastomosis. Dis Colon Rectum. 2003 Jan;46(1):20-3. doi: 10.1007/s10350-004-6491-7. PMID 12544517
- [Background] Madden MV, McIntyre AS, Nicholls RJ. Double-blind crossover trial of metronidazole versus placebo in chronic unremitting pouchitis. Dig Dis Sci. 1994 Jun;39(6):1193-6. doi: 10.1007/BF02093783. PMID 8200250
- [Background] Shen B, Achkar JP, Lashner BA, Ormsby AH, Remzi FH, Brzezinski A, Bevins CL, Bambrick ML, Seidner DL, Fazio VW. A randomized clinical trial of ciprofloxacin and metronidazole to treat acute pouchitis. Inflamm Bowel Dis. 2001 Nov;7(4):301-5. doi: 10.1097/00054725-200111000-00004. PMID 11720319
- [Background] Sambuelli A, Boerr L, Negreira S, Gil A, Camartino G, Huernos S, Kogan Z, Cabanne A, Graziano A, Peredo H, Doldan I, Gonzalez O, Sugai E, Lumi M, Bai JC. Budesonide enema in pouchitis--a double-blind, double-dummy, controlled trial. Aliment Pharmacol Ther. 2002 Jan;16(1):27-34. doi: 10.1046/j.1365-2036.2002.01139.x. PMID 11856075
- [Background] Mimura T, Rizzello F, Helwig U, Poggioli G, Schreiber S, Talbot IC, Nicholls RJ, Gionchetti P, Campieri M, Kamm MA. Four-week open-label trial of metronidazole and ciprofloxacin for the treatment of recurrent or refractory pouchitis. Aliment Pharmacol Ther. 2002 May;16(5):909-17. doi: 10.1046/j.1365-2036.2002.01203.x. PMID 11966499
- [Background] Nygaard K, Bergan T, Bjorneklett A, Hoverstad T, Lassen J, Aase S. Topical metronidazole treatment in pouchitis. Scand J Gastroenterol. 1994 May;29(5):462-7. doi: 10.3109/00365529409096839. PMID 8036463
- [Background] Gionchetti P, Rizzello F, Venturi A, Brigidi P, Matteuzzi D, Bazzocchi G, Poggioli G, Miglioli M, Campieri M. Oral bacteriotherapy as maintenance treatment in patients with chronic pouchitis: a double-blind, placebo-controlled trial. Gastroenterology. 2000 Aug;119(2):305-9. doi: 10.1053/gast.2000.9370. PMID 10930365
- [Background] Mimura T, Rizzello F, Helwig U, Poggioli G, Schreiber S, Talbot IC, Nicholls RJ, Gionchetti P, Campieri M, Kamm MA. Once daily high dose probiotic therapy (VSL#3) for maintaining remission in recurrent or refractory pouchitis. Gut. 2004 Jan;53(1):108-14. doi: 10.1136/gut.53.1.108. PMID 14684584
- [Background] Gionchetti P, Rizzello F, Helwig U, Venturi A, Lammers KM, Brigidi P, Vitali B, Poggioli G, Miglioli M, Campieri M. Prophylaxis of pouchitis onset with probiotic therapy: a double-blind, placebo-controlled trial. Gastroenterology. 2003 May;124(5):1202-9. doi: 10.1016/s0016-5085(03)00171-9. PMID 12730861
- [Background] Shen B, Brzezinski A, Fazio VW, Remzi FH, Achkar JP, Bennett AE, Sherman K, Lashner BA. Maintenance therapy with a probiotic in antibiotic-dependent pouchitis: experience in clinical practice. Aliment Pharmacol Ther. 2005 Oct 15;22(8):721-8. doi: 10.1111/j.1365-2036.2005.02642.x. PMID 16197493
- [Background] Chopra A, Pardi DS, Loftus EV Jr, Tremaine WJ, Egan LJ, Faubion WA, Hanson KA, Johnson TA, Sandborn WJ. Budesonide in the treatment of inflammatory bowel disease: the first year of experience in clinical practice. Inflamm Bowel Dis. 2006 Jan;12(1):29-32. doi: 10.1097/01.mib.0000192323.82426.83. PMID 16374255
- [Background] Gionchetti P, Rizzello F, Morselli C, et al. Eight-week trial of oral budesonide for the treatment of refractory pouchitis. Gastroenterology 126:A123, 2004
- [Background] Miglioli M, Barbara L, Di Febo G, Gozzetti G, Lauri A, Paganelli GM, Poggioli G, Santucci R. Topical administration of 5-aminosalicylic acid: a therapeutic proposal for the treatment of pouchitis. N Engl J Med. 1989 Jan 26;320(4):257. doi: 10.1056/NEJM198901263200423. No abstract available. PMID 2911318
- [Background] Viscido A, Habib FI, Kohn A, Papi C, Marcheggiano A, Pimpo MT, Vernia P, Cadau G, Caprilli R. Infliximab in refractory pouchitis complicated by fistulae following ileo-anal pouch for ulcerative colitis. Aliment Pharmacol Ther. 2003 May 15;17(10):1263-71. doi: 10.1046/j.1365-2036.2003.01535.x. PMID 12755839
- [Background] Gionchetti P, Rizzello F, Venturi A, Ferretti M, Brignola C, Peruzzo S, Belloli C, Poggioli G, Miglioli M, Campieri M. Long-term efficacy of bismuth carbomer enemas in patients with treatment-resistant chronic pouchitis. Aliment Pharmacol Ther. 1997 Aug;11(4):673-8. doi: 10.1046/j.1365-2036.1997.00217.x. PMID 9305474
- [Background] Tremaine WJ, Sandborn WJ, Kenan ML. Bismuth subsalicylate tablets for chronic antibiotic-resistant pouchitis. Gastroenterology 114:A1101, 1998.
- [Background] Wischmeyer P, Pemberton JH, Phillips SF. Chronic pouchitis after ileal pouch-anal anastomosis: responses to butyrate and glutamine suppositories in a pilot study. Mayo Clin Proc. 1993 Oct;68(10):978-81. doi: 10.1016/s0025-6196(12)62270-8. PMID 8412364
- [Background] Tremaine WJ, Sandborn WJ, Wolff BG, Carpenter HA, Zinsmeister AR, Metzger PP. Bismuth carbomer foam enemas for active chronic pouchitis: a randomized, double-blind, placebo-controlled trial. Aliment Pharmacol Ther. 1997 Dec;11(6):1041-6. doi: 10.1046/j.1365-2036.1997.00253.x. PMID 9663827